CLINICAL TRIAL: NCT01215955
Title: Two Approaches to Escalate Lispro Therapy in Patients With Type 2 Diabetes Mellitus Not Achieving Adequate Glycemic Control on Basal Insulin Therapy and Oral Agents Alone (AUTONOMY)
Brief Title: Study of Insulin Lispro in Participants With Inadequately Controlled Type 2 Diabetes
Acronym: AUTONOMY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13460; F3Z-MC-IOQC (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-09-30; First posted 2010-10-07 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Insulin; Algorithms; Blood glucose levels
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 Day Algorithm (Experimental): Basal insulin glargine plus mealtime bolus insulin lispro titrated based on blood glucose readings from the past three days.
  (Sites were assigned to Study A and Study B according to an allocation plan that was pre-specified before initiation of Study A and Study B)
  Interventions: Drug: Insulin lispro; Drug: Glargine
- Daily Algorithm (Experimental): Basal insulin glargine plus mealtime bolus insulin lispro titrated based on blood glucose readings from the previous day.
  (Sites were assigned to Study A and Study B according to an allocation plan that was pre-specified before initiation of Study A and Study B)
  Interventions: Drug: Insulin lispro; Drug: Glargine

INTERVENTIONS:
Drug: Insulin lispro — Administered subcutaneously, up to three times daily for 24 weeks
  Other Names: Humalog; LY275585
Drug: Glargine — Administered subcutaneously, dosage determined by investigator once daily for 24 weeks

SUMMARY:
Evidence regarding optimal methods of insulin dose adjustment is lacking in the literature. The purpose of this study is to evaluate the efficacy and safety of two approaches to escalate prandial insulin therapy in participants with type 2 diabetes mellitus not achieving adequate glycemic control on basal insulin.

DETAILED DESCRIPTION:
Participants who enter the study and are already taking insulin glargine with a screening HbA1c >7.0% will be randomized to one of two treatment arms. Both arms will add prandial insulin to existing basal insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Have been treated for at least 90 days with insulin glargine, neutral protamine Hagedorn (NPH), or detemir in combination with oral antihyperglycemic agents as monotherapy, dual, or triple therapy [sulfonylurea, meglitinide, metformin, pioglitazone, or dipeptidyl peptidase-4 (DPP-4) inhibitor] and in the opinion of the investigator requires further intensification of therapy
* Are treated with insulin glargine, NPH, or detemir at least 20 units per day (U/day) at enrollment
* Have an glycated hemoglobin (HbA1c) value greater than 7.0% and less than or equal to 12.0% according to the central laboratory at screening
* Capable of and willing to do the following: inject insulin with a prefilled pen, perform self blood glucose monitoring and record keeping as required by this protocol, as determined by the investigator
* Have given written informed consent to participate in this study in accordance with local regulations

Exclusion Criteria:

* Prior rapid- or short-acting insulin therapy: participants receiving scheduled long-term short-acting or rapid-acting or premixed insulin therapy within the past 6 months will not be eligible to participate in the study. Participants who have previously received short- or rapid-acting insulin as part of short-term insulin therapy (during gestational diabetes, during an acute hospitalization or illness) or occasional use will be allowed to participate in this study. Occasional use (e.g., used to treat acute hyperglycemia) shall be defined as less than daily administration of not more than 1 dose per day of short- or rapid-acting insulin
* Concomitant medications: glucagon-like peptide-1 (GLP-1) receptor agonist, alpha-glucosidase inhibitor, or rosiglitazone use concurrently or within 3 months prior to entry into the study
* Severe hypoglycemia: have had more than one episode of severe hypoglycemia (defined as requiring assistance of a third party due to disabling hypoglycemia) within 6 months prior to entry into the study
* Excessive insulin resistance: received a total daily dose of insulin greater than 2.0 units per kilogram (U/kg) at the time of randomization
* Morbid obesity: defined as a body mass index greater than or equal to 45 kilograms per square meter (kg/m²)
* Malignancy: have active or untreated malignancy, or have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer) for less than 5 years
* Cardiovascular: have cardiac disease with functional status that is New York Heart Association Class III or IV (see New York Heart Association Cardiac Disease Classifications) or have Congestive Heart Failure (CHF) requiring pharmacologic treatment or, in the investigator's opinion, have severe dependent edema (i.e., edema of the feet or ankles) or have any condition associated with hypoperfusion, hypoxemia, dehydration, or sepsis
* Renal: have a history of renal transplantation or are currently receiving renal dialysis or have serum creatinine greater than or equal to 2 milligrams per deciliter (mg/dL) if not on metformin
* Hepatic: have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) greater than 3 times the upper limit of the reference range as defined by the central laboratory
* Hematologic: have known hemoglobinopathy or chronic anemia or other known blood disorder
* Reproductive:(for women) are pregnant or intend to become pregnant during the course of the study; are sexually active women of childbearing potential not actively practicing birth control by a method determined by the investigator to be medically acceptable; or are breastfeeding
* Allergy: have known allergy to insulin lispro, insulin glargine, or excipients contained in these products
* Glucocorticoid therapy: receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 weeks immediately before screening
* Adherence to protocol: have any other condition (including known drug or alcohol abuse or psychiatric disorder) that precludes the participant from following and completing the protocol
* Prior participation: are currently enrolled in, or have participated in, an interventional medical, surgical, or pharmaceutical drug or device or off-label use study (an investigational study in which a medical or surgical treatment was given) within 30 days prior to entry into the study, or persons who have previously completed or withdrawn from this study (after having signed the informed consent document). Participants may be ineligible if they are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Non-approved drug: have been treated with a drug within the last 30 days that has not received regulatory approval at the time of study entry

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1117 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (76):
- United States (33):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewiston, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clarkson Valley, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flemington, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaver, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belém
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maringá
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottetown, Prince Edward Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Croatia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Slavonski Brod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Denmark (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frederiksberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolding
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bourges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Bouëxière
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
- Lithuania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raseiniai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ukmerge
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuauhtémoc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara Jalisco
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
- Puerto Rico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
- South Africa (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halfway House
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol had 2 independent studies (Study A, Study B) from which data was analyzed separately and independently: Participants were randomized to 1of the 2 treatment arms (Q1D, Q3D) at the site level. Sites were assigned to a study according to an allocation plan that was pre-specified before initiation of the study.
Groups:
- Study A Q1D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated dose was based on blood glucose reading from the previous day (Q1D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q1D at the site level: sites were assigned to Study A according to an allocation plan that was pre-specified before initiation of Study A.
- Study A Q3D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated dose was based on blood glucose readings from the past 3 days (Q3D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q3D at the site level: sites were assigned to Study A according to an allocation plan that was pre-specified before initiation of Study A.
- Study B Q1D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated dose was based on blood glucose reading from the previous day (Q1D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q1D at the site level: sites were assigned to Study B according to an allocation plan that was pre-specified before initiation of Study B.
- Study B Q3D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated dose was based on blood glucose readings from the past 3 days (Q3D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q3D at the site level: sites were assigned to Study B according to an allocation plan that was pre-specified before initiation of Study B.
Period: Overall Study
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Started | 268 | 263 | 292 (Three (3) participants from 1 site were excluded due to quality issues and validity of data.) | 294 (Two (2) participants from 1 site were excluded due to quality issues and validity of the data.)
Received at Least 1 Dose of Study Drug | 267 | 261 | 288 | 290
Completed | 223 | 210 | 244 | 241
Not Completed | 45 | 53 | 48 | 53
Not completed — Adverse Event | 1 | 4 | 2 | 3
Not completed — Death | 2 | 0 | 1 | 3
Not completed — Entry Criteria Not Met | 1 | 3 | 4 | 7
Not completed — Lack of Efficacy | 1 | 2 | 1 | 0
Not completed — Lost to Follow-up | 4 | 4 | 8 | 9
Not completed — Physician Decision | 4 | 10 | 8 | 11
Not completed — Protocol Violation | 17 | 13 | 8 | 8
Not completed — Sponsor Decision | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 14 | 15 | 13 | 9
Not completed — Quality Issues | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set-all participants who entered this study, completed the lead-in period (if applicable), were randomized and received ≥1 dose of study insulin, except the participants from the site excluded due to quality issues and data validity.
Groups:
- Study A Q3D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated based dose was on blood glucose readings from the past 3 days (Q3D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q3D at the site level: sites were assigned to Study A according to an allocation plan that was pre-specified before initiation of Study A.
- Total: Total of all reporting groups
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D | Total
Number analyzed (Participants) | 267 | 261 | 288 | 290 | 1106
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.89 (10.25) | 58.82 (9.46) | 57.71 (9.71) | 57.01 (10.61) | 57.83 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 138 | 155 | 155 | 581
  Male | 134 | 123 | 133 | 135 | 525
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100 | 96 | 91 | 95 | 382
  Not Hispanic or Latino | 150 | 153 | 182 | 177 | 662
  Unknown or Not Reported | 17 | 12 | 15 | 18 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 22 | 20 | 11 | 11 | 64
  Asian | 4 | 4 | 8 | 2 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 2
  Black or African American | 20 | 15 | 35 | 29 | 99
  White | 219 | 218 | 228 | 240 | 905
  More than one race | 1 | 2 | 4 | 6 | 13
  Unknown or Not Reported | 1 | 0 | 2 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Argentina | 28 | 28 | 37 | 38 | 131
  Austria | 0 | 1 | 4 | 1 | 6
  Brazil | 2 | 4 | 11 | 14 | 31
  Canada | 5 | 6 | 7 | 11 | 29
  Croatia | 3 | 3 | 4 | 5 | 15
  Denmark | 5 | 0 | 1 | 0 | 6
  France | 3 | 0 | 1 | 3 | 7
  Lithuania | 2 | 4 | 4 | 5 | 15
  Mexico | 31 | 31 | 21 | 25 | 108
  Poland | 9 | 8 | 15 | 15 | 47
  Puerto Rico | 26 | 19 | 7 | 7 | 59
  Romania | 9 | 6 | 11 | 10 | 36
  Russian Federation | 12 | 13 | 15 | 16 | 56
  South Africa | 1 | 2 | 11 | 13 | 27
  United States | 131 | 136 | 139 | 127 | 533

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Week Endpoint in Glycated Hemoglobin (HbA1c)
Description: The change from baseline to 24 weeks in the percentage of HbA1c in plasma. The Least Squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included the independent variables: fixed effects for treatment, country, sulfonylurea/meglitinide use, visit, treatment by visit interaction with baseline HbA1c as a covariate.
Time Frame: Baseline, 24 weeks
Population: Full Analysis Set: All participants who completed the lead-in period (if applicable), were randomized, received ≥1 dose of study insulin with a baseline value for HbA1C, except participants from the excluded site.
Measure: Least Squares Mean (Standard Error); unit: percentage HbA1c
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 267 | 261 | 288 | 290
percentage HbA1c | -1.00 (0.08) | -0.96 (0.08) | -0.98 (0.07) | -0.92 (0.07)
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; LS Mean Difference = 0.04, 95% CI 2-sided [-0.15 to 0.22] — No imputation was performed. Participants without a 24-week value were handled by the statistical model
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; LS Mean Difference = 0.06, 95% CI 2-sided [-0.12 to 0.24] — No imputation was performed. Participants without a 24-week value were handled by the statistical model

2. Secondary Outcome: Percentage of Participants Achieving Glycated Hemoglobin (HbA1c) Target Values
Description: Percentage of participants who achieved HbA1c levels of ≤7.0% or ≤6.5%.
Time Frame: 24-week endpoint
Population: Full Analysis Set: all participants who completed the lead-in period (if applicable), were randomized, received ≥1 dose of study insulin, except participants from the excluded site; last observation carried forward (LOCF) was used.
Measure: Number; unit: percentage of participants
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 267 | 261 | 288 | 290
percentage of participants
  HbA1c ≤7.0% | 49.81 | 42.53 | 49.31 | 42.41
  HbA1c ≤6.5% | 26.22 | 23.37 | 25.00 | 22.76
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.128, Regression, Logistic — P-value is for HbA1c ≤7.0% at endpoint (LOCF). Logistic regression included treatment and effects for baseline stratification variables: baseline HbA1c (≤8% or >8%), country and sulfonylurea/meglitinide use. Comparison calculated as Q3D versus Q1D; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.520 to 1.09]
Statistical Analysis 2: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.625, Regression, Logistic — P-value is for HbA1c ≤6.5% at endpoint (LOCF). Logistic regression included treatment and effects for baseline stratification variables: baseline HbA1c (≤8% or >8%), country and sulfonylurea/meglitinide use. Comparison calculated as Q3D versus Q1D; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.580 to 1.39]
Statistical Analysis 3: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.162, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.53 to 1.11]
Statistical Analysis 4: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.723, Regression, Linear — [p-value comment as in outcome 2, analysis 2]; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.61 to 1.40]

3. Secondary Outcome: Percentage of Participants ≥65 Years of Age Achieving Glycated Hemoglobin (HbA1c) Target Concentration
Description: Percentage of participants ≥65 years of age achieving HbA1c target concentration of ≤7.0% or ≤6.5%.
Time Frame: 24-week endpoint
Population: A subset of the Full Analysis Set: all participants who completed the lead-in period (if applicable), were randomized, received ≥1 dose of study insulin and were ≥65 years of age, except participants from the excluded site. Last observation carried forward (LOCF) was used.
Measure: Number; unit: percentage of participants
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 65 | 69 | 56 | 65
percentage of participants
  HbA1c ≤7% | 58.46 | 57.97 | 67.86 | 46.15
  HbA1c ≤6.5% | 27.69 | 36.23 | 35.71 | 21.54
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.701, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.520 to 2.67]
Statistical Analysis 2: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.249, Regression, Logistic — [p-value comment as in outcome 2, analysis 2]; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.710 to 3.70]
Statistical Analysis 3: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.015, Regression, Logistic — P-value is for HbA1c ≤7% at endpoint (LOCF). Logistic regression included treatment and effects for baseline stratification variables: baseline HbA1c (≤8% or >8%), country and sulfonylurea/meglitinide use. Comparison calculated as Q3D versus Q1D; Included treatment and effects for baseline stratification variables: Baseline HbA1c (≤8% or >8%), country and sulfonylurea/meglitinide use; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.13 to 0.80]
Statistical Analysis 4: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.078, Regression, Logistic — [p-value comment as in outcome 2, analysis 2]; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.17 to 1.10]

4. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Body Weight
Description: Body weight was measured twice at each indicated visit and the average of the 2 measurements was used for analyses. Least Squares (LS) mean calculated using mixed model repeating measure (MMRM) analysis that included baseline, treatment, country, sulfonylurea/meglitinide use, baseline glycated hemoglobin (HbA1c) strata (≤8% and >8%), visit and treatment-by-visit interaction .
Time Frame: Baseline, 24-weeks
Population: Full Analysis Set: all participants who completed the lead-in period (if applicable), were randomized and received ≥1 dose of study insulin with a baseline body weight, except participants from the excluded site.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 267 | 261 | 288 | 290
kilograms (kg) | 2.15 (0.27) | 2.96 (0.28) | 2.47 (0.24) | 1.97 (0.24)
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis — No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Differences = 0.81, 95% CI 2-sided [0.17 to 1.46]
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.108, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; LS Mean Differences = -0.50, 95% CI 2-sided [-1.12 to 0.11]

5. Secondary Outcome: Time to Reach Glycated Hemoglobin (HbA1c) Target Values
Description: Percentage of participants is the number of participants who achieved HbA1c target values of ≤6.5% or ≤7.0% during the specified time period divided by the total number of participants who did not discontinue from the study but had not reached HbA1c target at the beginning of the specified post baseline time period (≤100 days and ≥101 days). Participants who did not experience an outcome before discontinuation or completion of the study were censored using the date of discontinuation. Participants who were lost to follow up the date of discontinuation were considered to be the date of last contact.
Time Frame: Baseline through 24 weeks
Population: Full Analysis Set: all participants who completed the lead-in period (if applicable), were randomized, received ≥1 dose of study insulin, except participants from the excluded site. Censored participants: Study A: ≤6.5% Q1D=186 and Q3D=197; Study A ≤7.0% Q1D=120 and Q3D=134; Study B: ≤6.5% Q1D=206 and Q3D=212, Study B ≤7.0% Q1D=135 and Q3D=152.
Measure: Number; unit: percentage of participants
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 267 | 261 | 288 | 290
percentage of participants
  HbA1c ≤6.5% Post-Baseline ≤100 days | 19.48 | 10.73 | 17.36 | 14.48
  HbA1c ≤6.5% ≥101 days post-baseline | 14.80 | 18.00 | 14.81 | 16.14
  HbA1c ≤7.0% Post-Baseline ≤100 days | 37.45 | 33.72 | 37.15 | 33.10
  HbA1c ≤7.0% ≥101 days post-baseline | 31.54 | 26.90 | 28.75 | 24.56
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.182, Regression, Cox — Comparison is calculated as Q3D versus Q1D; Cox Regression model with effects for treatment and baseline stratification variables (HbA1c, country, sulfonylurea/meglitinide use) was used; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.57 to 1.11]
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.460, Regression, Cox — Comparison is calculated as Q3D versus Q1D; [statistical method as in outcome 5, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.65 to 1.22]

6. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Fasting Glucose
Description: Least Squares (LS) mean calculated using mixed model repeating measure (MMRM) analysis that included baseline, treatment, country, sulfonylurea/meglitinide use, baseline glycated hemoglobin (HbA1c) strata (≤8% and >8%), visit and treatment-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Full Analysis Set: all participants who completed the lead-in period (if applicable), were randomized, received ≥1 dose of study insulin with baseline fasting glucose values, except participants from the excluded site.
Measure: Least Squares Mean (Standard Error); unit: millimoles/liter (mmoles/L)
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 267 | 261 | 287 | 290
millimoles/liter (mmoles/L) | 0.08 (0.22) | 0.37 (0.23) | -0.36 (0.21) | 0.45 (0.21)
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; LS Mean Differences = 0.29, 95% CI 2-sided [-0.19 to 0.77] — No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; LS Mean Differences = 0.81, 95% CI 2-sided [0.30 to 1.31] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Fasting Glucose in Participants ≥65 Years of Age
Description: as for outcome 6
Time Frame: Baseline, 24 weeks
Population: A subset of the Full Analysis Set: all participants who completed the lead-in period (if applicable), were randomized, received ≥1 dose of study insulin, who are ≥65 years of age with baseline fasting glucose values, except participants from the excluded site.
Measure: Least Squares Mean (Standard Error); unit: millimoles/liter (mmoles/L)
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 65 | 69 | 55 | 65
millimoles/liter (mmoles/L) | 0.42 (0.44) | 1.01 (0.46) | -0.18 (0.50) | 0.96 (0.46)
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.242, Mixed Models Analysis — Comparison is calculated as Q3D versus Q1D; LS Mean Differences = 0.59, 95% CI 2-sided [-0.40 to 1.58] — No imputation was performed. Participants without a 24-week value were handled by the statistical model
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.082, Mixed Models Analysis — Comparison is calculated as Q3D versus Q1D; LS Mean Differences = 1.13, 95% CI 2-sided [-0.15 to 2.41] — No imputation was performed. Participants without 24-week values were handled by the statistical model

8. Secondary Outcome: Change From Baseline to 24 Week Endpoint in 1,5-anhydroglucitol (1,5-AG)
Description: Least Squares (LS) mean calculated using mixed model repeating measure (MMRM) analysis that included baseline treatment, country, sulfonylurea/meglitinide use, baseline glycated hemoglobin (HbA1c) strata (≤8% and >8%), visit and treatment-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Full Analysis Set: all participants who completed the lead-in period (if applicable), were randomized, received ≥1 dose of study insulin with baseline 1,5-AG value, except participants from the excluded site.
Measure: Least Squares Mean (Standard Error); unit: microgram/milliliter (mcg/mL)
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 266 | 261 | 288 | 290
microgram/milliliter (mcg/mL) | 3.24 (0.35) | 3.09 (0.36) | 3.22 (0.32) | 2.95 (0.31)
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.723, Mixed Models Analysis — Comparison is calculated as Q3D versus Q1D; LS Mean Differences = -0.15, 95% CI 2-sided [-0.95 to 0.66] — No imputation was performed. Participants without a 24-week value were handled by the statistical model
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.495, Mixed Models Analysis — Comparison is calculated as Q3D versus Q1D; LS Mean Differences = -0.28, 95% CI 2-sided [-1.08 to 0.52] — No imputation was performed. Participants without a 24-week value were handled by the statistical model

9. Secondary Outcome: Change From Baseline to 24 Weeks in 7-Point Self-Monitored Blood Glucose (SMBG) Profile
Description: 7-Point Self-Monitored Blood Glucose profiles are measures of blood glucose concentration taken 7 time a day at the morning pre-meal, morning 2-hours (HR) postprandial (PP), midday pre-meal, midday 2-hours post-meal, evening pre-meal, bedtime and 0300 hour (3 am). Each participant took measures over any 3 days and the average was calculated for each of the 7 time points. Least Squares (LS) mean calculated using mixed model repeating measure (MMRM) analysis that included baseline, treatment, country, sulfonylurea/meglitinide use, baseline glycated hemoglobin (HbA1c) strata (≤8% and >8%), visit and treatment-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Full Analysis Set: all participants who completed the lead-in period (if applicable), were randomized, received ≥1 dose of study insulin and had values at baseline and the specified timepoint, except participants from the excluded site.
Measure: Least Squares Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 266 | 261 | 288 | 290
milligrams/deciliter (mg/dL)
  Morning Pre-Meal (215, 200, 214, 219) | -3.97 (3.02) | -0.65 (3.12) | -1.24 (2.22) | 0.85 (2.18)
  Morning 2-HR PP (208, 194, 202, 201) | -41.57 (3.74) | -42.28 (3.86) | -43.80 (2.94) | -39.42 (2.93)
  Midday Pre-Meal (214, 199, 213, 219) | -42.37 (3.07) | -40.94 (3.16) | 38.57 (2.59) | -32.35 (2.52)
  Midday 2-HR PP (207, 195, 201, 203) | -45.75 (3.95) | -49.23 (4.06) | -53.45 (3.35) | -50.38 (3.33)
  Evening Pre-Meal (214, 200, 214, 215) | -46.75 (3.60) | -43.38 (3.70) | -41.59 (3.27) | -35.94 (3.21)
  Bedtime (214, 200, 214, 216) | -60.61 (4.78) | -62.86 (4.91) | -54.71 (4.10) | -43.52 (4.00)
  0300 hour (3 am) (203, 192, 194, 193) | -26.33 (3.87) | -23.96 (3.98) | -22.40 (3.75) | -13.39 (3.71)
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.245, Mixed Models Analysis — P-value is for Morning Pre-meal. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = 3.32, 95% CI 2-sided [-2.28 to 8.93]
Statistical Analysis 2: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.842, Mixed Models Analysis — P-value is for Morning 2-HR PP. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = -0.71, 95% CI 2-sided [-7.71 to 6.29]
Statistical Analysis 3: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.626, Mixed Models Analysis — P-value is for Midday Pre-Meal. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = 1.42, 95% CI [-4.32 to 7.16]
Statistical Analysis 4: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.358, Mixed Models Analysis — P-value is for Midday 2-Hr PP. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = -3.48, 95% CI 2-sided [-10.91 to 3.95]
Statistical Analysis 5: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.322, Mixed Models Analysis — P-value is for Evening Pre-meal. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = 3.38, 95% CI 2-sided [-3.32 to 10.07]
Statistical Analysis 6: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.617, Mixed Models Analysis — P-value is for Bed Time. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = -2.25, 95% CI 2-sided [-11.08 to 6.58]
Statistical Analysis 7: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.519, Mixed Models Analysis — P-value is for 0300 hours. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = 2.37, 95% CI 2-sided [-4.86 to 9.60]
Statistical Analysis 8: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.415, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 2.10, 95% CI 2-sided [-2.96 to 7.15]
Statistical Analysis 9: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.198, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 2]; LS Mean Difference = 4.38, 95% CI 2-sided [-2.30 to 11.06]
Statistical Analysis 10: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 3]; LS Mean Difference = 6.22, 95% CI 2-sided [0.14 to 12.29]
Statistical Analysis 11: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.426, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 4]; LS Mean Difference = 3.07, 95% CI 2-sided [-4.50 to 10.64]
Statistical Analysis 12: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.140, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 5]; LS Mean Difference = 5.66, 95% CI 2-sided [-1.86 to 13.17]
Statistical Analysis 13: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 6]; LS Mean Difference = 11.18, 95% CI 2-sided [1.74 to 20.63]
Statistical Analysis 14: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.037, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 7]; LS Mean Difference = 9.01, 95% CI 2-sided [0.53 to 17.49]

10. Secondary Outcome: Daily Dose of Insulin: Total, Basal and Prandial (Bolus)
Description: Total insulin was the sum of basal insulin (glargine) that was required to manage normal daily blood fluctuations and prandial insulin that was taken at meal time. Least Squares (LS) mean calculated using mixed model repeating measure (MMRM) analysis that included baseline, treatment, country, sulfonylurea/meglitinide use, baseline glycated hemoglobin (HbA1c) strata (≤8% and >8%), visit and treatment-by-visit interaction.
Time Frame: 24 weeks
Population: Full Analysis Set: all participants who completed the lead-in period (if applicable), were randomized, received ≥1 dose of study insulin and with values in the specified category, except participants from the excluded site.
Measure: Least Squares Mean (Standard Error); unit: international units (IU)
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 267 | 261 | 288 | 290
international units (IU)
  Basal Insulin (223, 213, 243, 239) | 65.53 (1.41) | 66.67 (1.44) | 61.24 (1.16) | 62.33 (1.15)
  Prandial (Bolus) Insulin (226, 213, 244, 241) | 47.10 (2.82) | 53.81 (2.87) | 43.03 (2.69) | 48.40 (2.68)
  Total Insulin (227, 213, 244, 242) | 110.52 (3.32) | 119.38 (3.43) | 103.08 (3.53) | 109.13 (3.51)
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.543, Mixed Models Analysis — P-value is for basal insulin dose. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = 1.15, 95% CI 2-sided [-2.55 to 4.84]
Statistical Analysis 2: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.095, Mixed Models Analysis — P-value is for bolus insulin dose. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = 6.72, 95% CI 2-sided [-1.17 to 14.60]
Statistical Analysis 3: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.059, Mixed Models Analysis — P-value is for total insulin dose. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = 8.86, 95% CI 2-sided [-0.35 to 18.06]
Statistical Analysis 4: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.497, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]; LS Mean Difference = 1.09, 95% CI 2-sided [-2.05 to 4.23]
Statistical Analysis 5: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.156, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 2]; LS Mean Difference = 5.37, 95% CI 2-sided [-2.06 to 12.79]
Statistical Analysis 6: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.222, Mixed Models Analysis — P-value of for total insulin dose. No imputation was performed. Participants without a 24-week value were handled by the statistical model. Comparison is calculated as Q3D versus Q1D; LS Mean Difference = 6.05, 95% CI 2-sided [-3.67 to 15.76]

11. Secondary Outcome: Daily Dose of Insulin Per Kilogram of Body Weight: Total, Basal and Prandial (Bolus)
Description: Total insulin was the sum of basal insulin (glargine) that was required to manage normal daily blood fluctuations and prandial insulin that was taken at meal time. Total, basal and prandial amounts were then divided by the participant's body weight in kilograms (kg). Least Squares (LS) mean calculated using mixed model repeating measure (MMRM) analysis that included baseline, treatment, country, sulfonylurea/meglitinide use, baseline glycated hemoglobin (HbA1c) strata (≤8% and >8%), visit and treatment-by-visit interaction.
Time Frame: 24 weeks
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: international units/kilogram (IU/kg)
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 267 | 261 | 288 | 290
international units/kilogram (IU/kg)
  Basal Insulin Dose (223, 213, 243, 239) | 0.68 (0.01) | 0.70 (0.01) | 0.64 (0.01) | 0.66 (0.01)
  Bolus Insulin Dose (226, 213, 244, 241) | 0.48 (0.02) | 0.55 (0.03) | 0.44 (0.02) | 0.47 (0.02)
  Total Insulin Dose (227, 213, 244, 242) | 1.12 (0.03) | 1.22 (0.03) | 1.09 (0.03) | 1.14 (0.03)
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.442, LS Mean Difference — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.02 to 0.05]
Statistical Analysis 2: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.037, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 2]; LS Mean Difference = 0.07, 95% CI 2-sided [0.00 to 0.14]
Statistical Analysis 3: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 3]; LS Mean Difference = 0.10, 95% CI 2-sided [0.05 to 0.16]
Statistical Analysis 4: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.275, LS Mean Difference — [p-value comment as in outcome 10, analysis 1]; LS Mean Difference = 0.02, 95% CI 2-sided [-0.01 to 0.05]
Statistical Analysis 5: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.194, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 2]; LS Mean Difference = 0.03, 95% CI 2-sided [-0.02 to 0.08]
Statistical Analysis 6: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.245, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 3]; LS Mean Difference = 0.06, 95% CI 2-sided [-0.04 to 0.15]

12. Secondary Outcome: The Number of Participants With a Hypoglycemic Episode (Incidence)
Description: A hypoglycemic episode was defined as any time a participant felt they were experiencing a sign or symptom that was associated with hypoglycemia, or had a blood glucose level of ≤70 milligram per deciliter [mg/dL, ≤3.9 millimoles per liter (mmol/L)] even if it was not associated with signs, symptoms or treatment (consistent with current American Diabetes Association 2005 guidelines).
Time Frame: Randomization through 24 weeks overall
Population: All randomized participants except from the excluded site.
Measure: Number; unit: participants
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 268 | 263 | 289 | 292
participants | 231 | 218 | 238 | 231
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.435, Regression, Logistic — Comparison is calculated as Q3D versus Q1D
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.351, Regression, Logistic — Comparison is calculated as Q3D versus Q1D

13. Secondary Outcome: The Number of Participants ≥65 Years of Age With Hypoglycemic Episodes (Incidence)
Description: A hypoglycemic episode in participants ≥ 65 years of age was defined as any time a participant felt they were experiencing a sign or symptom that was associated with hypoglycemia, or had a blood glucose level of ≤70 milligram per deciliter [mg/dL, ≤3.9 millimoles per liter (mmol/L)] even if it was not associated with signs, symptoms or treatment (consistent with current American Diabetes Association 2005 guidelines).
Time Frame: Randomization through 24 weeks overall
Population: All randomized participants ≥65 years old except those from the excluded site.
Measure: Number; unit: participants
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 66 | 69 | 56 | 65
participants | 60 | 61 | 51 | 53
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.802, Regression, Logistic — Comparison is calculated as Q3D versus Q1D
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.205, Regression, Logistic — Comparison is calculated as Q3D versus Q1D

14. Secondary Outcome: The Rate of Hypoglycemic Episodes
Description: The hypoglycemia rate per 30 days was calculated as the number of hypoglycemic episodes reported divided by the number of days at risk times 30.
Time Frame: Randomization through 24 weeks overall
Population: All randomized participants except those from the excluded site.
Measure: Mean (Standard Deviation); unit: hypoglycemic episodes per 30 day period
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 268 | 263 | 289 | 292
hypoglycemic episodes per 30 day period | 3.15 (0.23) | 3.33 (0.25) | 3.18 (0.26) | 3.33 (0.27)
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.586, Negative Binomial Regression — Comparison is calculated as Q3D versus Q1D; Q3D vs Q1D Ratio of Negative Binomial = 1.06, 95% CI 2-sided [0.86 to 1.30]
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.689, Negative Binomial — Comparison is calculated as Q3D versus Q1D; Q3D vs Q1D Ratio Negative Binomial = 1.05, 95% CI 2-sided [0.84 to 1.30]

15. Secondary Outcome: Percentage of Participants With Severe Hypoglycemic Episodes
Description: Severe hypoglycemia is defined as an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. Plasma glucose measurements may not be available during such an event, but neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by low plasma glucose.
Time Frame: Randomization up to 24 weeks
Population: All randomized participants except those from the excluded site.
Measure: Number; unit: percentage of participants
Groups:
- Study B Q1D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated based on blood glucose reading from the previous day (Q1D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q1D at the site level: sites were assigned to Study B according to an allocation plan that was pre-specified before initiation of Study B.
- Study B Q3D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated based on blood glucose readings from the past 3 days (Q3D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q3D at the site level: sites were assigned to Study B according to an allocation plan that was pre-specified before initiation of Study B.
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Number analyzed (Participants) | 268 | 263 | 289 | 292
percentage of participants | 1.9 | 0.8 | 2.4 | 2.7
Statistical Analysis 1: Comparison: Study A Q1D vs Study A Q3D; Test type: Superiority or Other; p = 0.258, Regression, Logistic — Comparison is calculated as Q3D versus Q1D
Statistical Analysis 2: Comparison: Study B Q1D vs Study B Q3D; Test type: Superiority or Other; p = 0.856, Regression, Logistic — Comparison is calculated as Q3D versus Q1D

ADVERSE EVENTS:
Description: The number of participants at risk does not include 3 participants in Study B Q1D and 2 participants in Study B Q3D who were from the site excluded due to quality issues and data validity.
Groups:
- Study A Q1D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated based on blood glucose reading from the previous day (Q1D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q1D at the site level: sites were assigned to Study A according to an allocation plan that was pre-specified before initiation of Study A.
- Study A Q3D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated based on blood glucose readings from the past 3 days (Q3D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q3D at the site level: sites were assigned to Study A according to an allocation plan that was pre-specified before initiation of Study A.
- Study B Q3D: Insulin lispro administered subcutaneously, up to 3 times daily for 24 weeks. Mealtime bolus of insulin lispro self-titrated based on blood glucose reading from the previous day (Q1D).
  Glargine participant-dependent doses, administered subcutaneously once daily for 24 weeks.
  Participants were randomized to Q3D at the site level: sites were assigned to Study B according to an allocation plan that was pre-specified before initiation of Study B.
Arm/Group | Study A Q1D | Study A Q3D | Study B Q1D | Study B Q3D
Serious Adverse Events (participants affected / at risk) | 21/268 | 17/263 | 21/289 | 27/292
Other Adverse Events (participants affected / at risk) | 136/268 | 142/263 | 130/289 | 150/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Study A Q1D (N=268) | Study A Q3D (N=263) | Study B Q1D (N=289) | Study B Q3D (N=292)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — Event resulted in death in arm Study A Q1D
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rickettsiosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Event resulted in death in arm Study A Q1D
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase mb increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 2 (4) | 9 (10) | 8 (8)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Event resulted in death
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/135 (0) | 0/124 (0) | 0/134 (0) | 1/136 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/133 (0) | 0/139 (0) | 1/155 (1) | 0/156 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0/133 (0) | 0/139 (0) | 1/155 (1) | 0/156 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study A Q1D (N=268) | Study A Q3D (N=263) | Study B Q1D (N=289) | Study B Q3D (N=292)
Diabetic retinopathy (Eye disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 12 (13) | 6 (6) | 15 (16) | 13 (13)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (9) | 11 (11) | 8 (8)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (3) | 4 (4) | 2 (3)
Vomiting (Gastrointestinal disorders) | 6 (7) | 4 (4) | 9 (10) | 6 (6)
Chest pain (General disorders) | 1 (1) | 5 (6) | 1 (2) | 3 (3)
Fatigue (General disorders) | 4 (4) | 3 (3) | 1 (1) | 8 (8)
Influenza like illness (General disorders) | 5 (5) | 5 (9) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 5 (5) | 6 (6) | 3 (3)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 3 (3) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 6 (6) | 10 (11) | 4 (4) | 7 (7)
Ear infection (Infections and infestations) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2) | 5 (5) | 7 (7)
Gastroenteritis viral (Infections and infestations) | 6 (6) | 3 (3) | 1 (1) | 4 (4)
Influenza (Infections and infestations) | 6 (7) | 8 (8) | 9 (14) | 12 (13)
Nasopharyngitis (Infections and infestations) | 19 (23) | 19 (19) | 12 (15) | 12 (12)
Pharyngitis (Infections and infestations) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 3 (4) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 7 (7) | 8 (9) | 4 (4) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 7 (8) | 5 (6) | 10 (10)
Urinary tract infection (Infections and infestations) | 8 (8) | 7 (8) | 3 (3) | 7 (9)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Weight increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 5 (5)
Dyslipidaemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 5 (7) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 11 (11) | 6 (6)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 2 (2) | 1 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 2 (3) | 5 (6) | 4 (4)
Headache (Nervous system disorders) | 4 (5) | 9 (10) | 13 (15) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 4 (4) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 4 (4) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 4 (4) | 9 (9)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 3 (3) | 3 (3)
Cataract operation (Surgical and medical procedures) | 3 (5) | 0 (0) | 3 (3) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 8 (8) | 13 (13) | 1 (1) | 5 (5)

LIMITATIONS AND CAVEATS:
Five (5) randomized participants (3 Study B Q1D, 2 Study B Q3D) from 1 site were excluded from efficacy and safety analyses due to quality issues and validity of the data at that site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days